CLINICAL TRIAL: NCT00580892
Title: Optical Coherence Tomography of Airway and Pleural Disorders
Status: Withdrawn | Type: Observational
Why Stopped: Not a clinical trial study
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Matthew Brenner, M.D.,Department of Pulmonary and Critical Care Medicine, University of California, Irvine
Other Study IDs: 20064982
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Disorder of Pleura and Pleural Cavity
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Airway and Pleural Disorders: Optical Coherence Tomography imaging
  Interventions: Device: Optical Coherence Tomography imaging

INTERVENTIONS:
Device: Optical Coherence Tomography imaging — Optical Coherence Tomography imaging

SUMMARY:
The researcher can use Optical coherence tomography a near-infrared diode to emit light that can produce images of the specimen under investigation and provide information about tissue abnormalities without causing damage.

DETAILED DESCRIPTION:
The researcher can use Optical coherence tomography endoscopic imaging to improve diagnosis and treatment of airway and pleural malignancy. In the events of burn injury and smoke inhalation injury, the Optical coherence tomography can determine the change of the airway tissues and severity of airway injury.

During endoscopic procedure the lesions will be biopsied and prepared by standard histologic methods. The Optical coherence tomography endoscopic imaging can measured histologic of the tissue samples and compared to standard histologic examination. The Optical coherence tomography endoscopic imaging can measured the epithelial thickness and compared to visual inspection of the mucosa on bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 or older, male or female.
* Plans for bronchoscopic with possible biopsy procedures.

Exclusion Criteria:

* Age less than 18 years of age
* Not plan for bronchoscopic with possible biopsy procedures.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selcted from University of California Irvine Chao Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
histopathology | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brenner, M.D, Principal Investigator — Beckman Laser Institute
Locations (1):
- Pulmonary and Critical Care Medicine, Irvine, California, United States